CLINICAL TRIAL: NCT02548273
Title: Corneal Changes in Diabetics After Phacoemulsification
Status: Completed | Type: Observational
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, DR.NIRUBAN.G, Dr., Jawaharlal Institute of Postgraduate Medical Education & Research
Other Study IDs: IEC/SC/2012/4/159
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus
Keywords: Corneal endothelium; phacoemulsification
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetics: diabetics with cataract who opted for phacoemulsification surgery
- controls: non-diabetics with cataract who opted for phacoemulsification surgery (subjects without corneal opacity, PXF ,high myopia, uveitis)

SUMMARY:
This study aims to assess the corneal damage after phacoemulsification and to assess the factors causing it in diabetics in comparison with non-diabetics.

DETAILED DESCRIPTION:
Title:

Corneal changes in diabetics after phacoemulsification

Introduction:

Cataract is one of the common cause of reversible blindness. In diabetics, Age-related cataract occurs earlier and nuclear cataract is more common and tends to progress rapidly. True diabetic cataract is a rare condition usually occurring in young adults due to the osmotic over-hydration of the lens. Initially a large number of fluid vacuoles appear underneath the anterior and posterior capsules, which is soon followed by the appearance of bilateral snowflake-like white opacities in the cortex.

Diabetic hyperglycemia also inhibits the function of Na+ k+ ATPase activity thereby causing dysfunction of the corneal endothelial cell layer. The endothelial cell morphology is also abnormal in diabetics. Polymegathism and Pleomorphism are noted. The cornea is also found to be thicker in diabetics owing to the slower recovery of corneal edema.

Phacoemulsification with intraocular lens implantation is one of the most common surgical procedures performed for cataract surgery with a smaller incision, which decreases the tissue injury, reduces post-operative pain and inflammation, and provides a rapid refractive stabilization. Surgeries that are done for cataract result in decrease in the endothelial count of which phacoemulsification has lesser degree of endothelial damage compared to those of other surgeries. Parameters like nucleus density(1), axial length(2) and the ultrasound power(3) also influence the endothelial cell count after phacoemulsification.

Aims and objectives:

1. To assess the central corneal thickness and endothelium after phacoemulsification in diabetics in comparison with non-diabetics.
2. To assess the factors associated with Corneal endothelial cell damage after phacoemulsification in diabetics in comparison with non-diabetics.

Review of literature:

Shultz et al(4) in the study on morphologic changes in corneal endothelial cells in diabetics for a duration of more than 21 years, found that diabetic corneal endothelial cell changes are caused continuously even after ocular operations, because the diabetic cornea is unstable and vulnerable. They found annual rates of reduction in corneal endothelial cells were 2.5% per year in operated eyes having extracapsular cataract extraction and 0.3% to 0.5% in normal individuals, thus showing a higher reduction rate in the surgically treated eyes by 10 year analysis.

Furuse and coauthors(5) compared the morphologic changes in corneal endothelial cells after performing planned Extra capsular cataract extraction on 96 normal aged cataract patients and diabetic patients. They observed that there was no significant difference between the 2 groups in terms of the density of corneal endothelial cells, the co-efficient of variation in cell size, and the cell hexagonality until 12 months postoperatively.

Goebbels and spitznas(6) performed flurophotometry of the corneal endothelium before and 4 days, 3 weeks and 6 weeks after phacoemulsification and intraocular lens implantation and endothelial permeability was evaluated in the presence or absence of diabetes mellitus. Endothelial permeability did not differ between the diabetic and non diabetic groups before operation, markedly increased in both groups 4 days after operation and recovered 3 weeks after operation in the non diabetic group but 6 weeks after operation in the diabetic group. This result was consistent with delayed recovery of endothelial function in the cornea of diabetic patients after cataract surgery.

Lee et al(7) studied the effect of the severity of retinopathy on endothelial loss post phacoemulsification and found an increased loss of endothelial cells and increased coefficient of variation in patients with high risk proliferative diabetic retinopathy when compared with patients with non proliferative diabetic retinopathy or patients without diabetes.

Su et al(8) designed a population based cross sectional study including 3239 eyes and examined the relationship of diabetics and CCT. They found that diabetes is associated with greater CCT, independent of age, sex and IOP levels.

Inoue et al(9) investigated corneal endothelial structure and corneal thickness in 99 eyes with type 2 diabetes and 97 control eyes without diabetes. They found a decrease in cell density and an increase in coefficient of variation and concluded that the corneal endothelial cell structure was damaged.

Materials and methods:

Whether the study involves humans : Humans only or animals or both

Type of study : Case control study Number of groups : 2 groups. Group 1 - phacoemulsification in diabetics Group 2 - phacoemulsification in non-diabetics.

Sample size : 80 patients in each group. The sample size is estimated with an expected difference of 19 in corneal thickness at 5% level of significance and 80% power. The minimum sample size estimated was 70 in each group. The sample size is further modified with an expected drop out of 10%.

The protocol was approved by the Institute Ethical Committee. The study was done on patients attending ophthalmology outpatient services for visual ailments.Essential data such as name, age, sex and hospital number of patients enrolled were noted. The purpose and details of the study were explained to each subject and after obtaining informed consent, patients were recruited into the study.

Preoperatively, detailed ocular examination including visual acuity (using Snellen's chart or equivalent E optotypes), refraction, slit lamp examination, corneal endothelial count and morphology assessment (ECD, CV, hexagonality) using Konan noncon robo specular microscope (Model - NSP 9900) and corneal thickness using ultrasonic pachymeter were done for all patients planned for phacoemulsification surgery. Specular microscopy and pachymetry were measured by the same observer for all subjects. CCT was measured after topical anesthesia using one drop of proparacaine eye drops (0.5% w/v) and an average of three readings was noted.

Intraoperative mydriasis, phacoemulsification time and power were noted. Postoperatively, visual acuity, ocular inflammation scores, corneal thickness, CD, CV and hexagonality were measured on the first week, six weeks and three months. Ocular inflammation score was calculated based on the SUN (Standardization of uveitis nomenclature) working group grading scheme for anterior chamber cells.

Method of analysis:

Test for differences between groups in terms of demographic and clinical characteristics was done using the Chi-Square test for categorical variables. Independent student's t test or Mann Whitney's U test was used for comparing continuous variables. To identify the independent factors associated with the outcome, multiple logistic regression analysis was used. Preoperative versus postoperative modifications within the groups were verified using two-way repeated measures ANOVA. All statistical tests were carried out at 5% level of significance and p value < 0.05 was considered statistically significant. Data analysis was performed using SPSS (version 20.0, SPSS Inc.).

Hypothesis:

There is an Increase in central corneal thickness and decrease in corneal endothelial count after phacoemulsification surgery in diabetics in comparison to non-diabetics.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patients with age-related cataract planned for phacoemulsification.

Exclusion Criteria:

1. Patients undergoing cataract surgery (Other than phacoemulsification)
2. High myopia (> -6D)
3. Presence of corneal opacities
4. Presence of pseudoexfoliation
5. Presence of uveitis

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the Ophthalmology OPD, JIPMER
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
CHANGE FROM BASELINE IN CORNEAL ENDOTHELIAL CELL DENSITY AT 3 MONTHS | 3 MONTHS
CHANGE FROM BASELINE IN COEFFICIENT OF VARIATION OF CELL SIZE AT 3 MONTHS | 3 MONTHS
CHANGE FROM BASELINE IN CORNEAL ENDOTHELIAL CELL HEXAGONALITY AT 3 MONTHS | 3 MONTHS
  expressed as %
CHANGE FROM BASELINE IN CENTRAL CORNEAL THICKNESS AT 3 MONTHS | 3 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: NIRUBAN GANESAN, MBBS, MS, Principal Investigator — Jawaharlal Institute of Postgraduate Medical Education & Research